CLINICAL TRIAL: NCT00481689
Title: Prospective, Open-Label, Noncomparative, Multicenter Study to Evaluate the Efficacy and Safety of Ciprofloxacin Extended Release (Cipro XR) 1000 mg Tablets Given Once Daily for 7 to 14 Days in the Treatment of Patients 18 Years or Older With Complicated Urinary Tract Infections Caused by Pseudomonas Aeruginosa and Other Common Uropathogens
Brief Title: Study To Evaluate The Efficacy And Safety Of Ciprofloxacin Extended-Release (Cipro® XR) 1000 mg Tablets Given Once Daily For 7 To 14 Days In The Treatment Of Patients 18 Years Or Older With Complicated Urinary Tract Infections Caused By Pseudomonas Aeruginosa And Other Common Uropathogens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11490
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Urinary Tract Infections
Keywords: Cipro; Complicated UTI; Pseudomonas aeruginosa
MeSH Terms: conditions — Urinary Tract Infections; Pseudomonas Infections | interventions — Ciprofloxacin

INTERVENTIONS:
Drug: Cipro XR (Ciprofloxacin, BAYQ3939) — Active Ciprofloxacin XR ( 1000mg) given for 7 to 14 days

SUMMARY:
Researchers want to find out if a drug called Cipro® XR (ciprofloxacin extended-release) can help people with a complicated urinary tract infection caused by a kind of bacteria called Pseudomonas aeruginosa. The study doctor will give Cipro XR to some people to see if it is safe and works to treat complicated urinary tract infections caused by Pseudomonas aeruginosa. The study doctor will also gather information about using Cipro XR to treat complicated urinary tract infections caused by other bacteria. About 500 people with complicated urinary tract infections who are 18 years old and older will join this study. Cipro XR is approved by the U.S. Food and Drug Administration (FDA) for the treatment of complicated urinary tract infections and acute uncomplicated pyelonephritis (inflammation of the kidney). The dose of Cipro XR used in this study (1000 mg a day for 7 to 14 days), has been shown to be safe and effective. This study is being done to gather more information on using this dose of Cipro XR for complicated urinary tract infections caused by Pseudomonas aeruginosa, as well as by other bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women, 18 years of age or older with a suspected complicated urinary tract infection with an onset of symptoms 72 hours or less prior to study entry
* Patients must present with a least one sign or symptom of a lower UTI (dysuria, urgency, frequency, suprapubic pain) or for spinal cord injury patients if such symptoms are not present, at least one of the following: fever (T > 38º C or 100.4º F orally), onset of urinary incontinence, increased spasticity, autonomic hyperreflexia, increased sweating, or cloudy and odorous urine.
* Patients must have at least one of the underlying conditions

  * Indwelling urinary catheter or intermittent catheterization
  * 100 mL of residual urine after voiding
  * Neurogenic bladder
  * Obstruction due to nephrolithiasis, tumor or fibrosis
  * Urinary retention due to benign prostatic hypertrophy, bladder cancer or other urological anatomic abnormalities
  * Patients must have pyuria prior to enrollment (within 48 hours) defined as > 10 leukocytes/mm3 in unspun urine by hemocytometer or > 5 leukocytes/hpf in resuspended sediment of centrifuged urine
  * Patients must have one clean-catch, midstream urine culture or culture from catheter (obtained using sterile technique, not from a Foley bag) that was obtained within 48 hours of enrollment and had a positive results:

    1. Defined as >= 100000 CFU/mL (>= 10000 CFU/mL for S. saprophyticus) for a causative pathogen
    2. If more than 1 pathogen is identified, each should be present at a colony count >= 100000 CFU/mL (>= 10000 CFU/mL for S. saprophyticus) to be included in the analysis
    3. For catheterized patients two or more pathogens (>= 100000 CFU/mL) (>= 10000 CFU/mL for S. saprophyticus) isolated from a baseline urine culture will be considered contaminants unless simultaneous blood culture yields the same pathogen(s)
    4. The causative pathogen must be susceptible to ciprofloxacin on in vitro susceptibility testing
    5. Enrollment and start of treatment is permitted prior to the availability of the culture report

Exclusion Criteria:

* Have a history of allergy to quinolones
* Are unable to take or inability to tolerate oral medications
* History of prostatitis or epididymitis
* Have signs and symptoms of pyelonephritis [all of the following: fever (T>38° C/100.4° F orally), chills, and flank pain or costovertebral angle tenderness]
* Have an intractable infection requiring > 14 days of therapy
* Have an uncomplicated UTI
* Have a renal transplant
* Have ileal loops or vesico-ureteral reflux
* Have a ciprofloxacin-resistant pathogen upon urine or blood culture
* Have received systemic antimicrobial therapy within 48 hours prior to enrollment
* Have a neutrophil count <1000/mm3, CD4 < 200/mm3 or other conditions associated with significant depression in host defense; HIV testing is not mandatory
* Have a requirement for concomitant systemic antibacterial therapy with agents not specified in this protocol
* Have significant liver impairment (baseline SGOT or SGPT and/or total bilirubin greater than 3 times the upper limit of normal)
* Have significant renal impairment (serum creatinine > 3.0 mg/dl or creatinine clearance < 30 mL/min/1.73 m2)
* Have a history of tendinopathy associated with fluoroquinolones
* Are pregnant, nursing or in whom pregnancy cannot be excluded or unreliable contraception is being used
* Have been diagnosed with a rapidly fatal underlying disease (death expected within 6 months)
* Have a requirement for concomitant administration of sucralfate or divalent and trivalent cations such as iron or antacids containing magnesium, aluminum or calcium
* Have been previously enrolled in this clinical study
* Have been taking an investigational drug in the last 30 days
* Have a history of a UTI or bacteruria with a urinary pathogen resistant to a fluoroquinolone within 6 months prior to current UTI episode
* Any of the following signs of sepsis:
* Systolic blood pressure < 90mm or a decrease of > 40mm from baseline
* Hypothermia (T< 35.6°C, core)
* Unexplained metabolic acidosis (pH < 7.3 with BE >= 5mmol/L or elevated lactate level)
* PaO2 < 75 mm/Hg on room air or PaO2 /FIO2 ratio < 250
* Acute renal failure (urine output < 0.5mL/kg/h for >= 1h)
* DIC ( PTT, PT, or platelets < 1/2 baseline or < 100,000)
* Acute deterioration in mental state
* Hemodynamic state (CI > 4L/min/m2 + SVR < 800 dyn-sec/cm-5)15

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-05; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and efficacy of ciprofloxacin XR for treatment of subjects with complicated urinary tract infections caused by P. aeruginosa and other urinary pathogens. | 28-42 days after therapy

SECONDARY OUTCOMES:
Clinical response | TOC visit
Clinical response post- treatment | 28-42 days after therapy
Adverse Event collection | Until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- United States (33):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Cudahy, California
  - Fresno, California
  - La Mesa, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - Torrance, California
  - Waterbury, Connecticut
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Watertown, Massachusetts
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Reno, Nevada
  - East Orange, New Jersey
  - Albuquerque, New Mexico
  - Manhasset, New York
  - North Massapequa, New York
  - Troy, New York
  - Eugene, Oregon
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - San Antonio, Texas
  - Richmond, Virginia
  - Tacoma, Washington
  - Cheyenne, Wyoming